CLINICAL TRIAL: NCT03694158
Title: Effect of IL-4RαR576 Polymorphism on Response to Dupilumab in Asthma, a Genotype-stratified, Randomized, Placebo- Controlled Trial
Brief Title: Investigating Dupilumab's Effect in Asthma by Genotype
Acronym: IDEA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Regeneron Pharmaceuticals (Industry); HealthBeacon Plc (Industry); Merck Sharp & Dohme LLC (Industry); Sanofi (Industry)
Responsible Party: Principal Investigator, Wanda Phipatanakul, Professor of Pediatrics, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P00029072; U01AI143514 (NIH)
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: This is a genotype stratified, double-blind, randomized, placebo-controlled, parallel-group, phase IV clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, placebo controlled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Dupilumab (Dupixent®) administered subcutaneously every two weeks. An initial dose of 600 mg (two 300 mg injections) followed by 300 mg given every other week.
  Interventions: Drug: Dupilumab
- Placebo group (Placebo Comparator): Placebo (preparation, administration, packaging, and labeling all equivalent to the treatment) administered subcutaneously every two weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dupilumab — anti-IL4 receptor antagonist
  Other Names: Dupixent®
  Arms: Treatment group
Other: Placebo — Placebo for Dupilumab (packaged/administered the same as the active drug)
  Arms: Placebo group

SUMMARY:
The Goal of this study is to investigate if individuals ages 12 years and older, carrying the IL-4RαR576 gene variant, will have a greater response to therapy acting directly on the anti-IL-4R. This will be conducted by examining the effect of a 48 week therapy with dupilumab on the rate of asthma exacerbations.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled parallel-group phase 4 clinical trial.

Patients will be genotyped and categorized as those with: 1) the wild type allele (Q576/Q576), 2) heterozygous allele (Q576/R576), or 3) homozygous mutant allele (R576/R576); the genotype associated with more severe disease.

After a run-in period of 2-12 weeks to determine asthma control, subjects who fulfill all inclusion/exclusion criteria will be randomized to receive either subcutaneous Dupilumab or placebo (1:1 randomization allocation ratio).

This study addresses fundamental mechanisms by which the IL-4Rα-R576 variant drives the TH2/TH17 disease endotype and the influence of this variant on response to Dupilumab therapy. It brings together individuals with deep clinical and scientific expertise in allergic diseases, including epidemiology, genetics, inflammation, and tolerance mechanisms to investigate, in a coordinated strategy, the hypothesis that the IL-4Rα-R576 variant drives TH2/TH17 cell inflammation by subverting allergen-specific iTreg cells into TH17 cells. Asthmatics bearing this endotype will be particularly likely to favorably respond to Dupilumab therapy by virtue of its prevention of iTreg cell reprogramming into TH17-like cells, potentially leading to their long-term stability and potential for sustained immune tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 12 years and older
2. Ability to provide informed consent
3. Ability to perform pulmonary function tests
4. Female participants of childbearing potential must have a negative urine pregnancy test upon study entry
5. Female participants with reproductive potential must agree to use FDA-approved methods of birth control for the duration of the study2
6. Participant-reported physician or licensed medical practitioner diagnosis of asthma
7. Treatment with medium to high dose ICS (400 mcg to maximum of 2000 mcg per day of fluticasone propionate or equivalent) for at least 3 months with a stable dose ≥1 month prior to screening OR used a biologic medication for asthma within the past 8 weeks
8. History of asthma exacerbation in the past year

An exacerbation is an asthma attack for which a clinician prescribed a course of systemic (oral, IV, IM) steroids whether or not the patient took the steroids OR An increase of >50% of baseline inhaled corticosteroid dose for ≥3 days OR An unscheduled visit for acute asthma attack (licensed medical practitioner/nurse office, urgent care intervention, emergency department, or hospitalization)

Exclusion Criteria:

1. Chronic lung disease other than asthma, which may impair lung function
2. Current smoker or cessation of smoking ≤6 months prior to Visit 0 screening
3. Current use of any electronic (e) "vaping" device (e.g., e-cigarette, e-cig, mod, vape pen, JUUL, e-cigar, e-hookah, e-pipe, vape pods) or cessation ≤ 6 months prior to screening
4. Pregnant or breast feeding
5. Any other condition or abnormality that, in the opinion of the Principal Investigator, would compromise the safety of the patient or quality of data
6. Evidence that the participant or family may be unreliable or poorly adherent to their asthma treatment or study procedures
7. Planning to relocate away from the clinical center area before study completion
8. Currently participating in an investigational drug trial or participated in one within 30 days before screening
9. Currently being treated with immunosuppressive/immunomodulatory or other investigational agents or biologics for conditions other than asthma, or used a biologic for a non-asthma indication within the past 6 months
10. History of respiratory illness requiring antibiotics or systemic corticosteroids, including asthma exacerbations, within the past 4 weeks (evaluated at time of screening visit)
11. History of alcohol or illicit substance abuse within 6 months of screening
12. Neutropenia (<1,000/mm3) or thrombocytopenia (<100,000/mm3) or hemoglobin < 100 g/L (10 g/dL) or blood eosinophils > 1500/mm3 at screening
13. Administration of a live vaccine within 4 weeks of screening
14. Currently receiving allergen immunotherapy (food or aeroallergen) other than an established maintenance regimen implemented continuously for a minimum of 2 months. Individuals receiving aeroallergen immunotherapy must be willing to stay on it for the duration of the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The rate of asthma exacerbations | 48 week treatment period
  An exacerbation is an asthma attack for which a clinician prescribed a course of systemic steroids, whether or not the patient took the steroids.

SECONDARY OUTCOMES:
Change in pre-bronchodilator lung function | average of week 4,12, 24,36 and 48 week
  the change in pre-bronchodilator FEV1% predicted from baseline
Change in CASI score | average of 4,12, 24, 36, and 48 week
  The change in CASI score from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Phipatanakul, MD, MS, Principal Investigator — Boston Children's Hospital
Locations (6):
- United States (6):
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Montefiore Einstein Clinical Research Center, The Bronx, New York
  - MetroHealth System, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lai PS, Massoud AH, Xia M, Petty CR, Cunningham A, Chatila TA, Phipatanakul W. Gene-environment interaction between an IL4R variant and school endotoxin exposure contributes to asthma symptoms in inner-city children. J Allergy Clin Immunol. 2018 Feb;141(2):794-796.e3. doi: 10.1016/j.jaci.2017.08.023. Epub 2017 Sep 21. No abstract available. PMID 28943468
- [Background] Massoud AH, Charbonnier LM, Lopez D, Pellegrini M, Phipatanakul W, Chatila TA. An asthma-associated IL4R variant exacerbates airway inflammation by promoting conversion of regulatory T cells to TH17-like cells. Nat Med. 2016 Sep;22(9):1013-22. doi: 10.1038/nm.4147. Epub 2016 Aug 1. PMID 27479084